CLINICAL TRIAL: NCT00200473
Title: A Double-Blind, Multi-Center, Randomized, Placebo-Controlled, Parallel Group Study of the Effects of Nebivolol on Safety and Efficacy in Patients With Mild to Moderate Hypertension
Brief Title: A Study of the Safety and Efficacy of Nebivolol in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB305
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: Nebivolol; Hypertension; Beta-Blockers
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

INTERVENTIONS:
Drug: Nebivolol

SUMMARY:
A study to determine the safety, efficacy and superiority of nebivolol to placebo for the treatment of elevated blood pressure in patients with mild to moderate hypertension.

DETAILED DESCRIPTION:
This study was a multi-center, multi-national, randomized, double-blind, parallel group, placebo-controlled study of nebivolol over a range of doses in patients with mild to moderate hypertension. The study consisted of 2 phases: screening/washout/single-blind placebo run-in and 2) randomization/double-blind treatment. Patients had 7 scheduled clinic visits during the study.

ELIGIBILITY:
Inclusion Criteria:

* An average sitting diastolic blood pressure of greater then or equal to 95 mmHg and less then or equal to 109 mmHg at baseline

Exclusion Criteria:

* Recent myocardial infarction or stroke
* Secondary hypertension
* Contraindications to beta-blocker therapy or discontinuation of prior antihypertensive agents
* Pregnancy, nursing or women of childbearing age not using appropriate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2001-09; Study Completion 2003-03

PRIMARY OUTCOMES:
The change of the average sitting diastolic blood pressure (24 plus/or minus 2 hours post-previous morning's dose) taken at trough at the end of the treatment compared to baseline

SECONDARY OUTCOMES:
- The change of the average sitting, supine and standing systolic and diastolic blood pressure at trough and peak at end of treatment compared to baseline
- Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Betty S. Riggs, MD, MBA, Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Mylan Pharmaceuticals Inc., Morgantown, West Virginia, United States